CLINICAL TRIAL: NCT07158021
Title: Phase 2 Randomized Trial to Examine Ovarian Function Suppression for Breast Cancer (OFS)
Brief Title: Leuprolide and Goserelin for Ovarian Function Suppression in Pre- or Peri-menopausal Women With Breast Cancer, OFS Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2025.016; NCI-2025-03933 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00270281 (Other: University of Michigan)
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm I (leuprolide) (Experimental): Patients receive lower dose leuprolide IM on day 1 of each cycle. Cycles repeat every 28 days for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Drug: Leuprolide; Other: Questionnaire Administration
- Arm II (leuprolide) (Experimental): Patients receive higher dose leuprolide IM on day 1 of each cycle. Cycles repeat every 28 days for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Drug: Leuprolide; Other: Questionnaire Administration
- Arm III (goserelin) (Experimental): Patients receive goserelin SC on day 1 of each cycle. Cycles repeat every 28 days for up to 24 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Drug: Goserelin; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Drug: Goserelin — Given SC
  Other Names: ICI-118630
  Arms: Arm III (goserelin)
Drug: Leuprolide — Given IM
  Other Names: Leuprorelin
  Arms: Arm I (leuprolide); Arm II (leuprolide)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares leuprolide to goserelin for reducing estrogen production by the ovaries in pre- or peri-menopausal women with breast cancer. Estrogen can cause the growth of breast cancer cells. Both leuprolide and goserelin lower the amount of estrogen made by the body. This may help stop the growth of tumor cells that need estrogen to grow. This study compares lower dose leuprolide, higher dose leuprolide, and goserelin for their ability to suppress the function of the ovaries to produce estrogen. Both doses of leuprolide may be as safe, tolerable and/or effective as goserelin in suppressing ovarian function in pre- or peri-menopausal women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female subject aged ≥ 18 years
* Pre- or peri-menopausal patient, who had (1) menses within the 12 months prior to enrollment or (2) estradiol concentration above the postmenopausal range per institutional laboratory guidance within the 12 months prior to enrollment
* Planning to take GnRHa therapy in combination with oral endocrine therapy (tamoxifen, anastrozole, exemestane, or letrozole) for adjuvant treatment of stage 1-3 breast cancer or for treatment of metastatic breast cancer
* Not planning bilateral salpingo-oophorectomy during the 6-month study duration
* Completion of chemotherapy, if given. Concurrent use of trastuzumab, pertuzumab, bisphosphonate therapy, poly adenosine diphosphate-ribose polymerase (PARP) inhibitor therapy, cyclin D kinase 4/6 (CDK4/6) inhibitor, and/or phosphoinositide 3-kinase (PI3K) inhibitor therapy is permitted
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Prior bilateral salpingo-oophorectomy
* Known to be pregnant or breastfeeding (negative pregnancy test will be confirmed prior to study treatment initiation)
* Concomitant use of systemic or transdermal estrogen products
* Known allergy or hypersensitivity to goserelin or leuprolide, or any of the excipients in the medications
* Unable to take oral medications
* Any medical condition that would interfere with the absorption of endocrine therapy. Prior gastric bypass is permitted
* Patients with a prior or concurrent malignancy whose natural history or treatment, in the opinion of the treating investigator, has the potential to interfere with the safety or efficacy assessment of the investigational regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ultrasensitive estradiol concentration > 10 pg/ml | During the first 24 weeks of therapy
  Analyses will primarily be descriptive reporting the overall and by treatment group proportions of women with ultrasensitive estradiol concentration and the corresponding exact binomial 95% confidence intervals over the first 24 weeks of gonadotropin releasing hormone agonist (GnRHa) therapy.

SECONDARY OUTCOMES:
Proportion of participants with ultrasensitive estradiol concentration > 10 pg/ml | At 4 weeks after initial GnRHa treatment administration
  Will be described with corresponding 95% confidence intervals overall and by treatment group.
Proportion of participants with ultrasensitive estradiol concentration > 10 pg/ml | Any time after 4 weeks of initial GnRHa treatment administration, assessed cycle 3 day 1-cycle 7 day 1 (cycle length = 28 days)
  Will be described with corresponding 95% confidence intervals overall and by treatment group.
Change in Functional Assessment of Cancer Therapy-(FACT)-Endocrine Subscale (ES) Trial Outcome Index | Up to 24 weeks
  Will use linear mixed-effects models with fixed effects for study group, time, and their interaction. For each outcome, a random intercept for each participant will be included to account for within-subject correlation. This approach allows for estimation of longitudinal trends in FACT-ES scores and assessment of whether changes over time differ between treatment arms. Missing data will be handled using maximum likelihood estimation under the assumption of missing at random (MAR).
Change in FACT-ES Endocrine Symptom Subscale | Up to 24 weeks
  Will use linear mixed-effects models with fixed effects for study group, time, and their interaction. For each outcome, a random intercept for each participant will be included to account for within-subject correlation. This approach allows for estimation of longitudinal trends in FACT-ES scores and assessment of whether changes over time differ between treatment arms. Missing data will be handled using maximum likelihood estimation under the assumption of MAR.
Percentage of participants reporting discomfort of 6/10 or higher on the Discomfort of Injection questionnaire | At the day following initial GnRHa injection
  Will be described by study arm and with corresponding exact binomial 95% confidence intervals.
Percentage of participants reporting discomfort of 6/10 or higher on the Discomfort of Injection questionnaire | Before administration of the second GnRHa injection
  Will be described by study arm and with corresponding exact binomial 95% confidence intervals.
Receipt of GnRHa therapy within ± 1 day of planned dosing | Up to 24 weeks
  Planned dosing should be given every 28 days. The proportion of patients who receive GnRHa therapy within ± 1 day of planned dosing will be reported overall and by study arm with corresponding exact binomial 95% confidence intervals.
Incidence of adverse events (AEs) | Up to 24 weeks
  AEs will be graded and described using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will be reported using descriptive statistics for each GnRHa study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
participant demographics, estradiol concentrations, and patient-reported outcomes data will be available to researchers upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: researchers can request data once the primary analysis has been published
Access Criteria: deidentified data will be available to researchers upon reasonable request